CLINICAL TRIAL: NCT00001393
Title: Genetic Markers for Focal Segmental Glomerulosclerosis
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940133; 94-DK-0133
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12-12

CONDITIONS: Focal Segmental Glomerulosclerosis; HIV-Associated Focal Segmental Glomerulosclerosis
Keywords: Collapsing Glomerulopathy; Renal Diseases; HIV-associated nephropathy; Natural History
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Kidney Diseases; AIDS-Associated Nephropathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- African descent controls: Controls; adult healthy volunteers of African descent without kidney disease
- African-Americans with FSGS: African-American patients with idiopathic or HIV-associated collapsing glomerulopathy
- African-Americans with HIV: Hyper-normal controls; adult African-Americans with HIV and without kidney disease
- European and Asian descent controls: Controls; healthy volunteers of European or Asian descent without kidney disease
- Kidney donors: People donating kidneys at NIH
- Other patients with idiopathic FSGS: Patients of other areas of descent with idiopathic FSGS
- Relatives of patients with familial FSGS: Relatives of patients with familial FSGS
- Tamils: Adults with Tamilian descent

SUMMARY:
Glomerulonephritis is a disease which affect the kidneys. Occasionally these diseases can progress to a loss of kidney function in some patients. Glomerulosclerosis or focal segmental glomerulosclerosis (FSGS) is one form of glomerulonephritis.

The cause of FSGS is unknown and often occurs on its own (idiopathic), or it can be associated with HIV (Human Immunodeficiency Virus). FSGS occurs more commonly among black patients than Caucasian or Hispanic patients. Researchers believe that environmental factors may interact with genetic mutations to cause FSGS, at least in some patients.

This study will attempt to identify genetic factors associated with the development of FSGS. The study population will be made up of 600 total subjects divided into 3 groups. Group one will be 200 African-Americans with FSGS. Group two will be 200 African-Americans with HIV but without FSGS. Group three will be 200 non-African-Americans with FSGS.

Study participation requires that researchers obtain 20 ml (2 tubes of blood). The genetic material (DNA) will be prepared from the white blood cells and analyzed. The results of each group will be compared with the results from the other groups to determine if one or more genes predisposes to FSGS. In the long run, studies that demonstrate a genetic basis for FSGS may help us identify patients earlier and may lead to improved therapies.

DETAILED DESCRIPTION:
Focal segmental glomerulosclerosis (FSGS) and a related condition, collapsing glomerulopathy, are chronic renal diseases affecting the glomerular podocytes. Currently, over thirteen genetic mutations are associated with FSGS. We are interested in expanding our understanding of these and other genes that may cause FSGS and collapsing glomerulopathy. We will study individuals with affected family members. We will also study sporadic cases; the rationale for studying this population is that FSGS and collapsing glomerulopathy are significantly more common among individuals of African descent. The latter observation suggests that particular FSGS-susceptibility alleles may be more common among African Americans. In the present study, we are addressing the hypothesis that genetic variation contributes to the pathogenesis of idiopathic FSGS and collapsing glomerulopathy, both idiopathic and HIV-associated variants. We are studying the following groups: 1) African-Americans with idiopathic or HIV-associated collapsing glomerulopathy. We will exclude post-adaptive FSGS, associated with glomerular hyperfiltration, and medication associated FSGS. 2) Other patients with idiopathic FSGS. 3) African Americans with HIV and without kidney disease (hyper-normal controls). 4) African descent controls (controls). 5) Healthy European and Asian descent controls (controls). 6) Relatives of patients with familial FSGS. 7) Kidney donors. 8) Tamils. We are taking four methodologic approaches. First, we are examining known FSGS risk genes or candidate genes, looking for disease-causing mutations and for disease-susceptibility haplotypes. Second, we have undertaken a genome scan, in the African descent population. We may also undertake a whole genome scan in European and Asian descent. Evidence of linkage disequilibrium among these markers will be sought between patients with and without FSGS. Third, when we identify families with multiple affected individuals and which lack known genetic mutations affecting FSGS genes, we will pursue positional cloning. Fourth, we will generate iPSC from peripheral blood from individuals with kidney disease (with a particular focus on those with particular genetic variants associated with glomerular disease) and from healthy volunteers. We will generate podocytes, to understand mechanisms of FSGS, and possibly macrophages, to understand reverse cholesterol transport (with relevance to nephrotic syndrome and more broadly cardiovascular disease).

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA, BY GROUP:

  1. African-descent with FSGS: renal biopsy showing FSGS or collapsing glomerulopathy, including HIV-associated collapsing glomerulopathy (HIV-associated nephropathy). We will include adult and pediatric patients. We will exclude patients with hyperfiltration FSGS.
  2. Other patients with FSGS (similar inclusion and exclusion criteria as in group 1).
  3. African descent with HIV and without kidney disease (controls). We will include adult patients who have had serologically confirmed HIV-1 infection for at least 8 years and lack clinical renal disease, as evidenced by normal creatinine and urine protein/creatinine ratio <0.5 or 24 hour urine protein excretion <500 mg/d.
  4. African descent (controls). We will include adults only. Exclusions will include HIV-1 infection, cardiovascular disease, and renal disease.
  5. European and Asian descent (controls). These samples represent DNA already obtained by Dr. Winkler s group under IRB approved protocols and these patients will not be recruited as part of the present study.<TAB>
  6. Relatives of patients with FSGS. In selected families (in which a patient has been found to have a mutation in an FSGS risk gene whose pathologic role has not been established), we will obtain individual histories of renal disease (hematuria, proteinuria, hypertension, nephrolithiasis) and will measure serum creatinine and urine protein excretion. We will include adults with and without renal disease and children with renal disease. We will evaluate children <18 years by obtaining a urine sample; if urinalysis and urine protein excretion are normal, we will not request a blood sample unless blood is being obtained for a clinical indication.
  7. Kidney donors. We will include NIH kidney donors only. We will obtain individual histories that provide information as to age, sex, race, surgical and medical histories, and family history. Our purpose is to examine whether particular genetic variants, including those in MYH9, influence the ability of the kidney to undergo hypertrophy following renal donation or the propensity to manifest albuminuria as a sign of glomerular stress. These findings have the potential to extend our understanding of the biology of MYH9 and might have clinical relevance for selecting kidney donors.
  8. Tamil population. We will recruit from a Tamil population. A Tamil will be defined as anyone that identifies themselves, their parents and their grandparents as Tamilian. We will ask these patients about their family history. We will exclude subjects under 18 and multiple subjects within the same family. We will draw blood for genetic testing. Our purpose is to determine whether particular genetic variants, including those in MYH9, are prevalent in a Tamilian population. If prevalence is indicated, we hope to study how these variants influence the progression of kidney disease in this population.
  9. Women who are pregnant will be excluded from participating in the apheresis component of this protocol.

Min Age: 19 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes several distinct populations of FSGS patients and healthy controls: patients of African descent, patients of Tamilian descent, healthy participants of African, European, Asian, and Tamilian descent, as well as people of African descent with HIV but without FSGS and adults who donate kidneys at NIH. The purpose of collecting samples for genetic analyses from these groups is to discover genetic variations that could be associated with FSGS, which is especially prevalent in African-American and Tamil populations.
Sampling Method: Non-Probability Sample
Enrollment: 616 (Actual)
Dates: Start 1996-04-15 (Actual)

PRIMARY OUTCOMES:
To develop a molecular understanding of racial differences in the incidence of podocyte diseases. | Retrospective and Prospective
  Addressing the hypothesis that genetic variation contributes to the pathogenesis of idiopathic FSGS and collapsing glomerulopathy, both idiopathic and HIV-associated variants.

CONTACTS AND LOCATIONS:
Overall Officials: Anirban Ganguli, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1994-DK-0133.html